CLINICAL TRIAL: NCT03565458
Title: An Open-label, Randomized, Multiple-dose, Crossover Study to Evaluate Drug-drug Interaction Following Oral Administration of Gemigliptin and Dapagliflozin or Empagliflozin in Healthy Adult Volunteers
Brief Title: Gemigliptin, Dapagliflozin, Empagliflozin DDI Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LG-DPCL018
Record Dates: First submitted 2018-05-24; First posted 2018-06-21 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — LC15-0444; dapagliflozin; empagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- gemigliptin (Experimental): gemigliptin single dose
  Interventions: Drug: Gemigliptin
- dapagliflozin (Experimental): dapagliflozin single dose
  Interventions: Drug: Dapagliflozin
- gemigliptin and dapagliflozin (Experimental): co-administration of gemigliptin and dapagliflozin
  Interventions: Drug: Gemigliptin; Drug: Dapagliflozin
- empagliflozin (Experimental): empagliflozin single dose
  Interventions: Drug: Empagliflozin
- gemigliptin and empagliflozin (Experimental): co-administration of gemigliptin and empagliflozin
  Interventions: Drug: Gemigliptin; Drug: Empagliflozin

INTERVENTIONS:
Drug: Gemigliptin — zemiglo 50mg,LG Chem
  Other Names: zemiglo
  Arms: gemigliptin; gemigliptin and dapagliflozin; gemigliptin and empagliflozin
Drug: Dapagliflozin — forxiga, dapagliflozin 10mg
  Other Names: forxiga
  Arms: dapagliflozin; gemigliptin and dapagliflozin
Drug: Empagliflozin — jardiance 25mg, empagliflozin
  Other Names: jardiance
  Arms: empagliflozin; gemigliptin and empagliflozin

SUMMARY:
gemigliptin,SGLT-2i DDI study

DETAILED DESCRIPTION:
LG-DPCL018 (gemigliptin,SGLT-2i DDI study) is to evaluate the safety and immunogenicity of gemilgliptin & dapagliflozin and gemigliptin & empagliflozin.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male adults at age between 19 to 55 at the time of the screening
2. Those whose BMI measurement result at screening visit is between 18 and 27 kg/m2
3. Subject who has voluntarily decided to participate in this clinical trial and consented after listening all procedures and objects of this clinical trial
4. subjects who is consented in writing to be sure to comply with the requirements of the clinical trial

Exclusion Criteria:

1. Subject who has past or present history of a clinically significant disease such as hepatic, renal, immunological, respiratory, musculoskeletal, endocrine, neurological, hemato-oncological, or cardiovascular disorder
2. Subject showing hypersensitivity reaction or having a history of hypersensitivity reaction that is clinically significant to gemigliptin or dapagliflozin or empagliflozin ingredients, drugs that contain same class of ingredients or other drugs(DPP-4i, SGLT-2i).
3. Subject who had infection disease or serious injury within 21 days before the randomization
4. Subject with genetic problems such as galactose intolerance, Lapp lactose dehydrogenase deficiency or glucose-galactose uptake disorder
5. Subject who do not have a medically approved contraceptive during the period of the clinical trial, or who plan to provide sperm
6. Subject who have received a clinical trial drug or a bioequivalence study drug within 90 days of the random allocation
7. Those who have received a drug that can significantly affect the absorption, distribution, metabolism or excretion of the clinical trial drug within 30 days of randomization
8. Subject who had whole blood donation within 60 days or component blood donation within 30 days before the randomization
9. subject who drinks the average amount per week exceeding 140 g of alcohol
10. Subject whose daily average smoking amount exceeds 20 pieces per day
11. Average daily grapefruit juice intake exceeding 2 cups
12. Subject who had a systolic blood pressure less than 100 mmHg, greater than 150 mmHg, diastolic blood pressure less than 70 mmHg, or greater than 100 mmHg at the time of screening test
13. Subject with a glomerular filtration rate of less than 60 mL / min / 1.73m^2 calculated from serum creatinine values at the time of screening
14. Subject whose blood creatinine, AST, ALT or γ-GT levels exceeded the upper limit of the reference range by 1.5 times the screening test
15. Subject who do not show a negative response in the hepatitis B test, hepatitis C test, HIV test and syphilis test
16. Subject who are sensitive to the ingredients of Yellow No. 5 or have an allergy history
17. Subject who have clinically significant abnormalities in other clinical tests
18. Subject with clinically significant abnormal ECG findings
19. Subject who is considered to be unsuitable in conducting the clinical trial at the principal investigator's discretionary judgment

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2018-08-20 (Estimated); Study Completion 2018-12-22 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of gemigliptin, dapagliflozin, empagliflozin | day1, day6, day7 0, 0.5, 1,1.5,2,2.5,3,4,5,6,8,12,16,24 hours
  AUCτ
Peak Plasma Concentration (Cmax) of gemigliptin, dapagliflozin, empagliflozin | day1, day6, day7 0, 0.5, 1,1.5,2,2.5,3,4,5,6,8,12,16,24 hours
  Css,max

SECONDARY OUTCOMES:
tss,max of gemigliptin, dapagliflozin, empagliflozin | day1, day6, day7 0, 0.5, 1,1.5,2,2.5,3,4,5,6,8,12,16,24 hours
  tss,max
minimum blood plasma concentration of gemigliptin, dapagliflozin, empagliflozin | day1, day6, day7 0, 0.5, 1,1.5,2,2.5,3,4,5,6,8,12,16,24 hours
  Css,min
Area under the plasma concentration versus time curve (AUC) of gemigliptin metabolite | day1,day6,day7 0, 0.5, 1,1.5,2,2.5,3,4,5,6,8,12,16,24 hours
  AUCτ
Peak Plasma Concentration (Cmax)of gemigliptin metabolite | day1,day6,day7 0, 0.5, 1,1.5,2,2.5,3,4,5,6,8,12,16,24 hours
  Css,max
minimum blood plasma concentration(Css,min) of gemigliptin metabolite | day1,day6,day7 0, 0.5, 1,1.5,2,2.5,3,4,5,6,8,12,16,24 hours
  Css,min
metabolic ratio of gemigliptin | day1,day6,day7 0, 0.5, 1,1.5,2,2.5,3,4,5,6,8,12,16,24 hours
  metabolic ratio

CONTACTS AND LOCATIONS:
Overall Officials: jungryul kim, doctor, Principal Investigator — samsung seoul medical center
Locations (1):
- LG chem, Seoul, Gangseo-Gu, South Korea